CLINICAL TRIAL: NCT04672785
Title: Long-term Outcomes in Terms of Disability and Quality of Life for Patients Undergoing Posterior Cranial Fossa Craniectomy in the Context of Compressive Cerebellar Hematoma
Acronym: CHANCE
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.355; 2020-A02717-32 (Registry Identifier: IDRC)
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-04

CONDITIONS: Craniectomy; Quality of Life; Cerebellar Haematoma; Handicaps Physical; Handicap Mental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent a posterior fossa craniectomy for a cerebellar hematoma
  Interventions: Behavioral: SF36 questionary

INTERVENTIONS:
Behavioral: SF36 questionary — patients who underwent a posterior fossa craniectomy for a cerebellar hematoma at Grenoble University Hospital between 01/01/2010 and 01/01/2020 were enrolled in this study. The main objective is to assess the level of disability and the quality of life of patients who have had a posterior cranial fossa craniectomy.

SUMMARY:
Posterior cranial fossa craniectomy has been shown to improve patient survival. The level of autonomy, disability and quality of life of survivors has been little studied and still underresearched,.

In this context, an assessment of the level of disability and of the quality of life after performing a posterior craniectomy seems relevant.

DETAILED DESCRIPTION:
Investigators are carrying out a retrospective observational, single-center study, in three intensive care units in the Grenoble Hospital Center. Every patients who underwent a posterior fossa craniectomy for a cerebellar hematoma at Grenoble University Hospital between 01/01/2010 and 01/01/2020 were enrolled in this study. The main objective is to assess the level of disability and the quality of life of patients who have had a posterior cranial fossa craniectomy. The primary outcome is the mRS(Modified Rankin score) measured at least one year following the ICU discharge. Secondary outcomes are the mRS(Modified Rankin Score) measured at discharge from the rehabilitation department, the GOS (Glasgow Outcome score) measured at least one year following the discharge from intensive care, and the SF36 (The Short Form 36)from the medical outcome study, score assessing the quality of life, collected via phone call.

ELIGIBILITY:
Inclusion Criteria:

* Patient who underwent a posterior cranial fossa craniectomy in the context of an acute cerebellar hematoma between January 01, 2012 to January 01, 2020.
* Adult man or woman
* Hospitalized in intensive care
* No opposition from the patient or a loved one to a telephone contact to determine the SF36 (The Short Form) quality of life scale, from the medical outcome study.

Exclusion Criteria:

* Subject under guardianship or subject deprived of liberty
* Early limitation of active therapy before 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patients who underwent a posterior fossa craniectomy for a cerebellar hematoma at Grenoble University Hospital between 01/01/2010 and 01/01/2020
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the level of handicap | through study completion, an average of 1 years post admission
  The mRS (Modified Ranking score) measured at least one year following the ICU discharge during the consultation after hospitalization in the medical file

SECONDARY OUTCOMES:
Global quality of life score | from january 2020, during 6 months
  the SF36 score assessing the quality of life, collected via phone call.
Neurological recovery | from january 2020, during 6 months
  the GOS (Glasgow Outcome Scale) score measured at least one year following the discharge from intensive care. It goes from 1 to 5.
  1 corresponds to death 5.Good Recovery

CONTACTS AND LOCATIONS:
Locations (1):
- CHUGA, Grenoble, France

IPD SHARING:
Plan to Share IPD: No